CLINICAL TRIAL: NCT02595723
Title: Phenytoin for Memory Impairment Secondary to Megestrol
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: The Rogosin Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 032015-004
Record Dates: First submitted 2015-07-02; First posted 2015-11-03 (Estimated); Results first posted 2019-09-09 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Phenytoin; Megestrol; Fluid Therapy

STUDY DESIGN:
Intervention Model Description: Each participant receives three treatments: phenytoin + megestrol, placebo + megestrol, or placebo + placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Phenytoin, Then Megestrol (Experimental): Participants first received pretreatment with Phenytoin 200 mg capsule twice/day for one day. Participants then received both Phenytoin (200 mg capsule twice/day) and liquid Megestrol (800 mg/day) for three consecutive days.
  Interventions: Drug: Phenytoin 200 mg capsule; Drug: Megestrol 800 mg liquid
- Placebo, Then Megestrol (Experimental): Participants first received pretreatment with Placebo (matching Phenytoin 200 mg capsule) twice/day for one day. Participants then received both Placebo (matching Phenytoin 200 mg capsule) twice/day and liquid Megestrol (800 mg/day) for three consecutive days.
  Interventions: Drug: Megestrol 800 mg liquid; Drug: Phenytoin-matched Placebo capsule
- Placebo, Then Placebo (Experimental): Participants first received pretreatment with Placebo (matching Phenytoin 200 mg capsule) twice/day for one day. Participants then received both Placebo (matching Phenytoin 200 mg capsule) twice/day and liquid Placebo (matching liquid Megestrol 800 mg/day) for three consecutive days.
  Interventions: Drug: Phenytoin-matched Placebo capsule; Drug: Megestrol-matched liquid Placebo

INTERVENTIONS:
Drug: Phenytoin 200 mg capsule — Phenytoin oral capsule was initiated on Day 1 and administered at 200 mg twice/day for four consecutive days (Days 1 - 4).
  Arms: Phenytoin, Then Megestrol
Drug: Megestrol 800 mg liquid — Liquid megestrol 800 mg/was initiated on Day 2 and administered at 09:00 for three consecutive days (Days 2 - 4).
  Arms: Phenytoin, Then Megestrol; Placebo, Then Megestrol
Drug: Phenytoin-matched Placebo capsule — Phenytoin-matched oral Placebo capsule was initiated on Day 1 and administered for four consecutive days (Days 1 - 4).
  Arms: Placebo, Then Megestrol; Placebo, Then Placebo
Drug: Megestrol-matched liquid Placebo — Megestrol-matched liquid placebo was initiated on Day 2 and administered at 09:00 for three consecutive days (Days 2 - 4).
  Arms: Placebo, Then Placebo

SUMMARY:
This study is designed to test if megestrol acetate induces changes in declarative memory in healthy controls and if pre-administration of phenytoin can ameliorate any induced cognitive impairments.

DETAILED DESCRIPTION:
Healthy adults (n=20) will be recruited and informed consent will be obtained. Participants will agree to a number of visits, a Baseline Visit, 6 Study Visits, and a follow-up Safety Visit. Each course of study drug will be followed by a washout, but allowed preexisting medications will not be stopped for study participation. A small subset (n=4) of participants will also undergo MRI scanning as a component of their visits following drug administration.

Baseline Visit: Cognition will be assessed by a variety of measures, which will determine baseline declarative memory and working memory. Mood will be assessed by a psychiatric interview, self-assessments, and a review of any standing physical symptoms will be completed for comparison to any side effects which develop after medication administration. Vital signs will be recorded and women will be screened for pregnancy. Blood will be collected for complete blood count (CBC) and comprehensive metabolic panel (CMP).

Visit 1: Participants will be randomized to one of three treatment possibilities: 1) phenytoin with megestrol, 2) placebo with megestrol, 3) placebo with placebo. Participants will receive phenytoin (200 mg BID) or placebo and will be instructed to take this medication for one full day (two doses) before starting their megestrol. They will take this medication for a total of 3.5 days.

Visit 2: After the participants have completed their medication course on the morning of this visit day, they will return to have cognition and mood reassessed. Vital signs will be taken and blood will be drawn to assess CMP, CBC, cortisol and phenytoin levels. Participants will now enter a "washout" period of this medicine combination (approximately 3 weeks) before returning for their next visit. For those participants offered the MRI scans, their visit will extend to approximately 3 hours.

Visit 3: Participants will return and be randomized to one of remaining two treatment possibilities as detailed above. Participants will again be instructed to start the first medication and take for one full day before taking the second medication, and will be instructed to take their second medication at starting the following day after starting the first medication at 0900 hours and continue taking the drugs for 3 consecutive days.

Visit 4: After the participants have completed their medication course on the morning of this visit day, they will return to have cognition and mood reassessed; completing all previously administered assessments excepting the Structured Clinical Interview for the Diagnostic and Statistical Manual of Mental Disorders (SCID). Vital signs will be taken and blood will be drawn to assess CMP, CBC, cortisol and phenytoin levels. Participants will now enter a "washout" period of this medicine combination (approximately 3 weeks) before returning for their next visit. For those participants offered the MRI scans, their visit will extend to approximately 3 hours.

Visit 5: Participants will return and receive the remaining treatment possibility, detailed above. Participants will again be instructed to start the first medication and take for one full day before taking the second medication and will be instructed to take their second medication at starting the following day after starting the first medication at 0900 hours and continue taking the drugs for 3 consecutive days.

Visit 6: After the participants have completed their medication course on the morning of this visit day, they will return to have cognition and mood reassessed. Vital signs will be taken and blood will be drawn to assess CMP, CBC, cortisol and phenytoin levels. Participants will now enter a "washout" period of this medicine combination (approximately 3 weeks) before returning for their final visit. For those participants offered the MRI scans, their visit will extend to approximately 3 hours.

Safety Visit: Participants will return for a final "safety" visit which will evaluate any remaining side effects, take vital signs, and include a final urinary pregnancy test (for women).

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women age 18-50 years
* Education of ≥ 12 years and baseline Rey Auditory Verbal Learning Test (RAVLT) total words recalled score ≥ 40 (normal baseline memory)
* Body mass index (BMI) between 18.5-35
* The ability to read and speak English as not all neurocognitive assessments have been translated and validated in other languages.

Exclusion Criteria:

* History (lifetime) of Bipolar Disorder, Major Depressive Disorder, psychotic depressive, schizophrenic, schizoaffective, or other Axis I psychotic disorders
* Has an unstable general medical condition (GMC) or significant medical condition, including but not limited to myocardial infarction, cancer, diabetes (hypertension is allowed if condition is being treated and is stable)
* Vulnerable populations including pregnant or nursing women, the incarcerated, or those with severe cognitive disorders
* Education history that includes Special Education or history of mental disability
* History of psychotropic medication therapy in the past 30 days
* Baseline Quick Inventory of Depressive Symptoms-Clinician Rated (QIDS-C) > 5
* Initiation of new medications within 14 days of the baseline visit, with the exception of over-the-counter (OTC) as needed medications (e.g. Tylenol, Advil, Motrin, etc.)
* Significant hypertensive blood pressure at baseline, defined as either systolic pressure > 150 or diastolic pressure > 95
* Febrile at baseline, defined as body temperature ≥ 100.5°F (38°C)
* Baseline heart rate > 100 bpm or < 50 bpm
* Medical history of diseases with central nervous system (CNS)-involvement, including but not limited to stroke, traumatic brain injury, and loss of consciousness > 1 minute
* History of allergic reaction or medical contraindication to megestrol or phenytoin
* Clinically significant abnormalities on baseline labs (e.g. hypokalemia, hypernatremia, anemia)
* Lifetime history of an immunosuppressive disorder or immunosuppressive therapy with within the past 6 months
* History of blood clots such as myocardial infarction (MI), stroke, deep vein thromboses (DVTs), pulmonary embolism (PE) or blood clotting disorder
* Currently actively suicidal or considered a high suicide risk (e.g. more than one lifetime suicide attempt or any attempt in the past 12 months)
* Any reason not listed which, as determined by the principle investigator (PI), would affect participant safety in the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2015-07; Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: E. Sherwood Brown, MD, PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 35 patients were screened for eligibility between July 2015 and September 2016.
Pre-assignment Details: 21 of 35 participants were randomized. Of those not randomized, 14 did not meet inclusion criteria.
Groups:
- Ph + Meg, Then Pl + Meg, Then Pl + Pl: Participants first received pretreatment with Phenytoin 200 mg capsule twice/day for one day. Participants then received both Phenytoin (200 mg capsule twice/day) and liquid Megestrol (800 mg/day) for three consecutive days.
  Following first 21-day washout, participants then received both Placebo (matching Phenytoin 200 mg capsule) twice/day and liquid Megestrol (800 mg/day) for three consecutive days.
  Following second 21-day washout, participants then received both Placebo (matching Phenytoin 200 mg capsule) twice/day and liquid Placebo (matching liquid Megestrol 800 mg/day) for three consecutive days.
- Pl + Meg, Then Pl + Pl, Then Ph + Meg: Participants first received pretreatment with Placebo (matching Phenytoin 200 mg capsule) twice/day for one day. Participants then received both Placebo (matching Phenytoin 200 mg capsule) twice/day and liquid Megestrol (800 mg/day) for three consecutive days.
  Following first 21-day washout, participants then received both Placebo (matching Phenytoin 200 mg capsule) twice/day and liquid Placebo (matching liquid Megestrol 800 mg/day) for three consecutive days.
  Following second 21-day washout, participants then received both Phenytoin (200 mg capsule twice/day) and liquid Megestrol (800 mg/day) for three consecutive days.
- Pl + Pl, Then Ph + Meg, Then Pl + Meg: Participants first received pretreatment with Placebo (matching Phenytoin 200 mg capsule) twice/day for one day. Participants then received both Placebo (matching Phenytoin 200 mg capsule) twice/day and liquid Placebo (matching liquid Megestrol 800 mg/day) for three consecutive days.
  Following first 21-day washout, participants then received both Phenytoin (200 mg capsule twice/day) and liquid Megestrol (800 mg/day) for three consecutive days.
  Following second 21-day washout, participants then received both Placebo (matching Phenytoin 200 mg capsule) twice/day and liquid Megestrol (800 mg/day) for three consecutive days.
Period: First Intervention (4 Days)
Arm/Group | Ph + Meg, Then Pl + Meg, Then Pl + Pl | Pl + Meg, Then Pl + Pl, Then Ph + Meg | Pl + Pl, Then Ph + Meg, Then Pl + Meg
Started | 8 | 6 | 7
Completed | 8 | 6 | 7
Not Completed | 0 | 0 | 0
Period: First Washout (21 Days)
Arm/Group | Ph + Meg, Then Pl + Meg, Then Pl + Pl | Pl + Meg, Then Pl + Pl, Then Ph + Meg | Pl + Pl, Then Ph + Meg, Then Pl + Meg
Started | 8 | 6 | 7
Completed | 6 | 6 | 7
Not Completed | 2 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Period: Second Intervention (4 Days)
Arm/Group | Ph + Meg, Then Pl + Meg, Then Pl + Pl | Pl + Meg, Then Pl + Pl, Then Ph + Meg | Pl + Pl, Then Ph + Meg, Then Pl + Meg
Started | 6 | 6 | 7
Completed | 6 | 6 | 7
Not Completed | 0 | 0 | 0
Period: Second Washout (21 Days)
Arm/Group | Ph + Meg, Then Pl + Meg, Then Pl + Pl | Pl + Meg, Then Pl + Pl, Then Ph + Meg | Pl + Pl, Then Ph + Meg, Then Pl + Meg
Started | 6 | 6 | 7
Completed | 6 | 5 | 7
Not Completed | 0 | 1 | 0
Period: Third Intervention (4 Days)
Arm/Group | Ph + Meg, Then Pl + Meg, Then Pl + Pl | Pl + Meg, Then Pl + Pl, Then Ph + Meg | Pl + Pl, Then Ph + Meg, Then Pl + Meg
Started | 6 | 5 | 7
Completed | 6 | 5 | 7
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ph + Meg, Then Pl + Meg, Then Pl + Pl | Pl + Meg, Then Pl + Pl, Then Ph + Meg | Pl + Pl, Then Ph + Meg, Then Pl + Meg | Total
Number analyzed (Participants) | 8 | 6 | 7 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.63 (3.97) | 30.50 (7.94) | 30.71 (9.20) | 29.48 (7.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 5 | 14
  Male | 3 | 2 | 2 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 2 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 2 | 5
  White | 4 | 3 | 5 | 12
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Rey Auditory Verbal Learning Test (RAVLT)
Description: Rey Auditory Verbal Learning Test (RAVLT) is a test of verbal learning and declarative memory. During the test, 15 nouns that are read aloud for 5 consecutive trials. Each trial is followed by a free recall test (participant is asked to recall the words that were just read to them). The sum of correctly recalled words across 5 trials is called the total raw score. The raw scores on the total recall (number of words correct across trials 1-5) are converted to standardized T-scores (Mean=50; SD=10; range 20-100) based on participant age and gender. The scores below are presented as T-scores, with higher scores indicative of better performance.
Time Frame: 4 days after intervention administration
Measure: Mean (Standard Deviation); unit: T-scores
Arm/Group | Phenytoin, Then Megestrol | Placebo, Then Megestrol | Placebo, Then Placebo
Number analyzed (Participants) | 20 | 19 | 19
T-scores | 51.89 (8.08) | 45.90 (10.40) | 48.37 (10.42)
Statistical Analysis 1: Comparison: Phenytoin, Then Megestrol vs Placebo, Then Megestrol vs Placebo, Then Placebo; Test type: Other; p = 0.003, Mixed Models Analysis — Overall group difference adjusted for prior group, time, and baseline values; Model includes prior group, time, and baseline values to control for possible effects

ADVERSE EVENTS:
Time Frame: 4 days for each intervention.
Description: The safety population included all participants who received at least one dose of intervention.
Arm/Group | Phenytoin, Then Megestrol | Placebo, Then Megestrol | Placebo, Then Placebo
All-Cause Mortality (participants affected / at risk) | 1/20 | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 5/20 | 0/19 | 5/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phenytoin, Then Megestrol (N=20) | Placebo, Then Megestrol (N=19) | Placebo, Then Placebo (N=19)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Transient hearing loss (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Mild cognitive impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Knee injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Irregular menses (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 2 (2)
Fall (Social circumstances) | 1 (1) | 0 (0) | 0 (0)
Cold (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No